CLINICAL TRIAL: NCT00342043
Title: Multidisciplinary Studies of Malaria Protection by Hemoglobinopathies and G6PD Deficiency in Mali
Brief Title: Examination of Protective Factors Against Severe Malaria
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905214; 05-I-N214
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-16

CONDITIONS: Malaria; Severe Malaria
Keywords: Sickle Trait; Fetal Hemoglobin; Hemoglobin C; Beta-Thalassemia; Artesunate-Amodiaquine
MeSH Terms: conditions — Malaria; beta-Thalassemia

SUMMARY:
This study, sponsored by the National Institutes of Health and the University of Bamako in Mali, Africa, will examine factors that may protect against progression of malaria from mild to severe disease. Infection with the malaria parasite causes disease ranging in severity from mild or no symptoms to severe. A better understanding of what factors protect against disease progression may help scientists develop improved methods of disease prevention and treatment. The objectives of this study are to:

* Identify differences in protective factors for severe malaria in Malinke children residing in two Mali villages, Kela and Kangaba. Genetic variations in hemoglobin proteins called HbS and HbC appear to confer protection against severe disease in some children but not others. HbC appears to protect young Malinke children living in Kela, but not in nearby Kangaba, while HbS protects children in Kangaba but not in Kela. In addition, deficiency of an enzyme produced by red blood cells called G6PD protects males, but not females, from severe malaria.
* Investigate how fetal hemoglobin (HbF) may protect against malaria in infants and determine how HbS, HbC, G6PD deficiency, and beta-thalassemia trait affect the rate of HbF decline during the first 2 years of life.

Children under 11 years of age who seek medical care at Kangaba or Kela health centers for symptoms of malaria may be eligible for this study. Each will be screened with a medical history, physical examination and blood test. In addition, healthy infants born to women referred to field site clinics may be enrolled for the newborn study. Participants undergo the following procedures:

Children with mild malaria are treated with artesunate and amodiaquine. Those with severe malaria are treated with quinine. Blood is collected by finger prick every day for 4 days to evaluate the response to treatment and for genetic testing. Some blood is stored for future research related to malaria.

Newborns have a heel or finger prick at 1, 3 and 6 months to collect a small blood sample for genetic testing. In addition, at the time of birth, a small amount of blood is collected from one of the blood vessels of the placenta. Some infants may be followed up to 2 years, with additional drops of blood taken at 12, 18 and 24 months. Some of the blood is stored for future research related to malaria.

DETAILED DESCRIPTION:
Our previous case-control study (protocol #01-I-N020) established that hemoglobin (Hb) C protects against severe malaria in the Dogon ethnic group of Mali, West Africa. We believe that abnormal display of major parasite virulence antigens (PfEMP-1) on the surface of HbC erythrocytes accounts for this protection. Whether this mechanism mediates protection by other mutant erythrocytes remains to be investigated. The principal objective of the current protocol has been to investigate whether HbC also protects against severe malaria in the Malinke of Kela, which historically gave rise to the Dogon. Our preliminary data from protocol #02-I-N285 suggest that HbC but not HbS (sickle trait) protects the young Malinke children of Kela, with the opposite being true for the Malinke children of Kangaba, a nearby village. To confirm these novel preliminary findings and to investigate candidate mechanisms of protection, our ongoing case-control study requires an additional 150 severe malaria patients who are less than 5 years old, of Malinke ethnicity, reside in either Kangaba or Kela villages, and have normal G6PD activity. Children less than 11 years old and diagnosed with either severe (case) or uncomplicated (control) malaria will be tested for hemoglobinopathies and G6PD deficiency. Severe and uncomplicated malaria patients will be treated with parenteral quinine or oral artemisinin combination therapies, respectively, which are standard of care in Mali. Principal outcome measures will include a comparison of the frequency of HbC, HbS, and G6PD deficiency between cases and controls; with odds ratios and 95% confidence intervals determining the degree and statistical significance of severe malaria protection.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. All malaria patients enrolled in the case-control study will be less than 11 years old.
  2. Uncomplicated malaria: Axillary temperature greater than 37.5 degrees Celsius or history of fever, signs and symptoms of malaria (e.g. headache, body aches, malaise), asexual parasite density less than 500,000 per microliter of blood, no criteria of severe malaria (see next paragraph), and no other etiologies of febrile illness (e.g. respiratory tract infection, cellulitis) on clinical examination.
  3. Severe malaria: Asexual parasite density greater than or equal to 100,000/uL or parasitemia of any density plus any one of the following: coma (defined as Blantyre coma score less than or equal to 2), convulsions (witnessed by investigator), severe prostration, severe anemia (hemoglobin less than 5 g/dL), respiratory distress, hypoglycemia (serum glucose less than 40 mg/dL), jaundice/icterus, shock (systolic blood pressure less than 50 mmHg, rapid pulse, cool extremities), cessation of eating and drinking, repetitive vomiting.

EXCLUSION CRITERIA:

Patients who are parasitemic yet are found by clinical examination to have another etiology of febrile illness (e.g., respiratory tract infection, cellulitis) will not be formally enrolled into the protocol, but may be treated for both malaria and their coexisting infection by the study team.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4850
Dates: Start 2005-08-02; Study Completion 2009-04-16

CONTACTS AND LOCATIONS:
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Agarwal A, Guindo A, Cissoko Y, Taylor JG, Coulibaly D, Kone A, Kayentao K, Djimde A, Plowe CV, Doumbo O, Wellems TE, Diallo D. Hemoglobin C associated with protection from severe malaria in the Dogon of Mali, a West African population with a low prevalence of hemoglobin S. Blood. 2000 Oct 1;96(7):2358-63. PMID 11001883
- [Background] Ayi K, Turrini F, Piga A, Arese P. Enhanced phagocytosis of ring-parasitized mutant erythrocytes: a common mechanism that may explain protection against falciparum malaria in sickle trait and beta-thalassemia trait. Blood. 2004 Nov 15;104(10):3364-71. doi: 10.1182/blood-2003-11-3820. Epub 2004 Jul 27. PMID 15280204
- [Background] Bard H. The postnatal decline of hemoglobin F synthesis in normal full-term infants. J Clin Invest. 1975 Feb;55(2):395-8. doi: 10.1172/JCI107943. PMID 1127106